CLINICAL TRIAL: NCT03447535
Title: Observational Study on Intrafamilial Oppositional Defiant Disorder (IODD) in Children and Adolescents
Brief Title: Better Understand Children and Adolescents' Intrafamilial Oppositional Defiant Disorder
Acronym: TOPi
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0443
Record Dates: First submitted 2018-02-02; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Oppositional Defiant Disorder With Familial Setting
Keywords: Oppositional defiant disorder; Family; Disruptive, impulse control and conduct disorders; Anxiety disorder; Intrafamilial disruptive behaviours disorder
MeSH Terms: conditions — Oppositional Defiant Disorder; Disruptive, Impulse Control, and Conduct Disorders; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- classic oppositional defiant disorder: CODD Group: " classic " oppositional defiant disorder
  SDQ total difficulties score and the parents report SDQ total difficulties score:
  Group CODD (" classic " oppositional defiant disorder): teacher report SDQ total difficulties score (≥ 12), parents report SDQ total difficulties score (≥14)
  Interventions: Other: Semi-directive interview (Kiddy Sads); Other: SDQ questionnaires (strenghs and difficulties questionnaire)
- intrafamilial oppositional defiant disorder: IODD group: intrafamilial oppositional defiant disorder
  SDQ total difficulties score and the parents report SDQ total difficulties score:
  Group IODD (Intrafamilial Oppositional Defiant Disorder): teacher report SDQ total difficulties score normal (<12), parents report SDQ total difficulties score abnormal (>16)
  Interventions: Other: Semi-directive interview (Kiddy Sads); Other: SDQ questionnaires (strenghs and difficulties questionnaire)

INTERVENTIONS:
Other: Semi-directive interview (Kiddy Sads) — semi-directive interview (Kiddy Sads) conducted as part of the care
Other: SDQ questionnaires (strenghs and difficulties questionnaire) — SDQ questionnaires (strenghs and difficulties questionnaire) conducted as part of the care

SUMMARY:
Oppositional Defiant Disorder (ODD) is defined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5) as: "A pattern of angry/irritable mood, argumentative/defiant behavior, or vindictiveness lasting at least 6 months exhibited during interaction with at least one individual who is not a sibling." "The disturbance in behavior is associated with distress in the individual or others in his or her immediate social context (e.g., family, peer group, work colleagues), or it impacts negatively on social, educational, occupational, or other important areas of functioning." Children with "classic" oppositional defiant disorder, except for mild forms, show symptoms in several settings (at home, at school, with peers).

In this study, the investigators will consider the specifics of children presenting "intrafamilial" oppositional defiant disorder (IODD). These children's symptoms are confined to only one setting: the home. Therefore, the aim of this study will be to characterize children with intrafamilial oppositional defiant disorder. The investigators want to understand the differences between IODD and classical forms of ODD in terms of psychiatric comorbidities, medical histories and cognitive abilities. They also investigate what clinicians currently do to help these families.

DETAILED DESCRIPTION:
Definition: Extended description of the protocol, including more technical information (as compared to the Brief Summary), if desired. Do not include the entire protocol; do not duplicate information recorded in other data elements, such as Eligibility Criteria or outcome measures.

Limit: 32,000 characters.

Child-to-parent violence was kept secret for a long time. Searchers don't know much about this type of domestic violence, however they recently tried to investigate more on the subject. Bousquet et al. carried out a review of literature on the subject, and grouped the articles that they found. There was only one study concerned with children with Intrafamilial Oppositional Defiant Disorder (IODD) which is called in the study Oppositional Defiant Disorder with family tyranny (Delaunay et al., 2008).

IODD is described in the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM) as a mild form of Oppositional Defiant Disorder (ODD). This term characterizes children that meet the criteria for ODD ("a pattern of angry/irritable mood, argumentative/defiant behavior, or vindictiveness") but their symptoms are confined to only one setting: the home. Therefore, the aim of this study is to characterize Intrafamilial ODD children and the particularities of their families.

Nowadays, new treatment strategies exist in Montpellier, designed to be used as group therapies. In these groups, non-violent resistance methods are taught to the parents. The efficiency of this therapy is currently being studied. To improve this therapy and to offer appropriate therapies to the children themselves, it is important to improve the acknowledgement of these "tyrannical children". This is the aim of this study. To reach this goal, the investigators will compare the medical records of the children with IODD to those of the children with classic ODD.

On one hand, they expect children with IODD to be more anxious and smarter than children with "classic" ODD. On the other hand, they expect they will have had diseases that changed interactions with their parents. They also assume they will come from small families: i.e. they may be an only child, educated by a single parent, or they may have wealthy parents. Finally, they hypothesize that clinicians won't treat the children with IODD the same way as those with "classic" ODD.

ELIGIBILITY:
Inclusion criteria:

* Child diagnosed with ODD with KSADS_PL
* Child who was evaluated during a day evaluation at one of our unit cares: UDS (Unité de Diagnostic et de Soins) or UPP (Unité de Prévention Pédosychiatrique)
* Child included in the "REACT" study
* 16 years old or under

Exclusion criteria:

* Child who has not been diagnosed with ODD
* Missing data in the parent report SDQ or teacher report SDQ preventing the SDQ total score calculation

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects include:
  * Patients diagnosed with ODD during a day evaluation at one of our unit cares: UDS (Unité de Diagnostic et de Soins) or UPP (Unité de Prévention Pédosychiatrique); both units are headed by the Pr Diane Purper-Ouakil CHU Saint Eloi Montpellier.
  * Patients included in the " REACT " study conducted at CHU Saint Eloi Montpellier, and diagnosed with ODD during the pre-study visit.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Measure of the prevalence of the anxiety disorder diagnosis | 1 day
  The psychometric test used to characterize the specific primary outcome measure is the Kiddie-SADS-PL Schedule For Affective Disorders and Schizophrenia for School Age Children Present and Lifetime Version.
  The K-SADS-PL is a semi-structured interview aimed at early diagnosis of affective disorders such as anxiety disorder, depression, bipolar disorder. It generates reliable and valid child psychiatric diagnoses (1). It is specifically designed for school children aged 6 to 18. In this study, the K-SADS-PL test is performed by psychiatry residents or by psychologists.
  The interview is performed during the evaluation day (hospital day care) or during the pre-study visit for patients participating in the " react " protocole.

SECONDARY OUTCOMES:
Measure of Intellectual qQuotient | 1 day
  The Wechsler Intelligence Scale for Children (WISC) is an individually administered intelligence test for children aged 6 to 16.
  The test generates a Full Scale IQ (formerly known as an intelligence quotient or IQ score) that represents a child's general intellectual ability.
  In our study, both WISC IV and WISC V have been used. The Fifth Edition is the most current version, and has therefore been used for the most recent tests.
  The WISC IV provides four index scores: Verbal Comprehension Index, Processing speed Index,Working Memory Index, Perceptual Reasoning Index (see below).
  The WISC V provides 5 index scores: Verbal Comprehension Index, Visual Spatial Index, Fluid Reasoning Index, Working Memory Index, and Processing Speed Index (see below).
  For the measure of the intellectual quotient and for the measure of all the index scores, the average is 80-120. Bellow average values represents poorer outcome.

OTHER OUTCOMES:
Assesment of Verbal Comprehension Index | 1 day
  The Verbal Comprehension Index (VCI) is a score derived from the administration of selected subtests from the fourth and the fifth Wechsler Intelligence Scale for Children (WISC). It is designed to provide a measure of verbal acquired knowledge and verbal reasoning. (See Encyclopedia of Clinical Neuropsychology)
Perceptual Reasoning Index | 1 day
  The WISC IV provides four index scores: Verbal Comprehension Index, Processing speed Index,Working Memory Index, Perceptual Reasoning Index.
  The WISC V provides 5 index scores: Verbal Comprehension Index, Visual Spatial Index, Fluid Reasoning Index, Working Memory Index, and Processing Speed Index.
Working Memory Index | 1 day
  The WISC IV provides four index scores: Verbal Comprehension Index, Processing speed Index,Working Memory Index, Perceptual Reasoning Index.
  The WISC V provides 5 index scores: Verbal Comprehension Index, Visual Spatial Index, Fluid Reasoning Index, Working Memory Index, and Processing Speed Index.
Processing Speed Index | 1 day
  The WISC IV provides four index scores: Verbal Comprehension Index, Processing speed Index,Working Memory Index, Perceptual Reasoning Index.
  The WISC V provides 5 index scores: Verbal Comprehension Index, Visual Spatial Index, Fluid Reasoning Index, Working Memory Index, and Processing Speed Index.
Visuo Spatial Index | 1 day
  The WISC IV provides four index scores: Verbal Comprehension Index, Processing speed Index,Working Memory Index, Perceptual Reasoning Index.
  The WISC V provides 5 index scores: Verbal Comprehension Index, Visual Spatial Index, Fluid Reasoning Index, Working Memory Index, and Processing Speed Index.
Fluid Reasoning Index (FRI) | 1 day
  It is a score derived from the administration of selected subtests from the fifth Wechsler Intelligence Scale for Children (WISC).
  It allows to detect underlying conceptual relationships among visual objects
Prevalence of somatic diseases in patient medical history | 1 day
  Past somatic diseases were mentioned in the patient medical record. We classified them into:
  1. Serious illness (chronic illness, hospitalisation needed, treatment taken for several months)
  2. Less serious illness.
Socio-economic status of the family assessed by parents' occupation | 1 day
  Parents' occupation were classified into 6 categories derived from the INSEE classification (Institut national de la statistique et des études économiques)
Family situation | 1 day
  Family situation: number of siblings, birth rank among siblings, single parents, divorced parents Description:This information is in the medical reports, it is mentioned in the questionnaire that is always filled by parents before the first consultation of their child.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa BOUSQUET, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC